CLINICAL TRIAL: NCT03261947
Title: An Open-Label, Phase 2, Parallel Arm Study to Evaluate the Safety, Tolerability, and Activity of TAK-931 Single Agent in Patients With Metastatic Pancreatic Cancer, Metastatic Colorectal Cancer, and Other Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, and Activity of TAK-931 in Participants With Metastatic Pancreatic Cancer, Metastatic Colorectal Cancer, and Other Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-931-2001; U1111-1192-7975 (Registry Identifier: World Health Organization); JapicCTI-163200 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Pancreatic Cancer; Colorectal Cancer; Esophageal Neoplasms; Carcinoma, Non-small-cell Lung
Keywords: Drug therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — simurosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Western Safety Cohort (Experimental): TAK-931 50 mg (2x25 mg or 5x10 mg), capsules, orally, once daily (QD) for 14 days, followed by a 7-day washout period (14 days on and 7 days off study drug), in 21-day cycles until disease progression or unacceptable treatment-related toxicity up to 20 cycles. Participants with locally advanced or metastatic solid tumors with no standard therapeutic alternative in the United States were included in this cohort.
  Interventions: Drug: TAK-931
- Pancreatic Cancer Cohort (Experimental): TAK-931 50 mg (2x25 mg or 5x10 mg), capsules, orally, QD for 14 days, followed by a 7-day washout period (14 days on and 7 days off study drug), in 21-day cycles until disease progression or unacceptable treatment-related toxicity up to 4 cycles. Participants with metastatic pancreatic cancer who had progressed after at least 1 line of standard chemotherapy were included in this cohort.
  Interventions: Drug: TAK-931
- Metastatic CRC Cohort (Experimental): TAK-931 50 mg (2x25 mg or 5x10 mg), capsules, orally, QD for 14 days, followed by a 7-day washout period (14 days on and 7 days off study drug), in 21-day cycles until disease progression or unacceptable treatment-related toxicity up to 12 cycles. Participants with metastatic CRC who had progressed after at least 2 lines of previous standard chemotherapy were included in this cohort.
  Interventions: Drug: TAK-931
- sqEC Cohort (Experimental): TAK-931 50 mg (2x25 mg or 5x10 mg), capsules, orally, QD for 14 days, followed by a 7-day washout period (14 days on and 7 days off study drug), in 21-day cycles until disease progression or unacceptable treatment-related toxicity up to 8 cycles. Participants with metastatic sqEC who had progressed after at least 1 line of standard chemotherapy were included in this cohort.
  Interventions: Drug: TAK-931
- sqNSCLC Cohort (Experimental): TAK-931 50 mg (2x25 mg or 5x10 mg), capsules, orally, QD for 14 days, followed by a 7-day washout period (14 days on and 7 days off study drug), in 21-day cycles until disease progression or unacceptable treatment-related toxicity up to 18 cycles. Participants with metastatic sqNSCLC who had progressed after at least 2 lines of standard treatment were included in this cohort.
  Interventions: Drug: TAK-931

INTERVENTIONS:
Drug: TAK-931 — TAK-931 hard gelatin capsules

SUMMARY:
The purpose of this study is to confirm the safety and tolerability of TAK-931 in a cohort of Western participants with metastatic solid tumors and to evaluate the anti-tumor activity of TAK-931 in participants with metastatic pancreatic cancer, colorectal cancer (CRC), squamous esophageal cancer (sqEC), and squamous non-small-cell lung cancer (sqNSCLC).

DETAILED DESCRIPTION:
Pancreatic Arm Now Closed.

The drug being tested in this study is called TAK-931. TAK-931 blocks function of a specific protein called CDC7 kinase in the human body. TAK-931 is being tested in participants with metastatic cancer (colorectal, pancreatic, sqNSCLC and sqEC) in the United States and Japan and also in the participants with any type of metastatic cancer with no standard therapeutic alternative in the United States only. This study will look at the safety, tolerability and pharmacokinetics of TAK-931.

The study will enroll approximately 160 participants. Participants will be enrolled in 5 cohorts: 1) Western safety cohort, to be enrolled in the United States only, will include non-Japanese participants with metastatic solid tumors and no standard therapeutic alternative, 2) Metastatic pancreatic cancer cohort, 3) Metastatic colorectal cancer cohort, 4) Metastatic sqNSCLC cohort, and 5) Metastatic sqEC cohort. All participants will receive:

• TAK-931 50 mg (2x25 mg or 5x10 mg) capsules

All participants will be asked to take one 50 mg (2x25 mg or 5x10 mg) capsule at the same time of the day every day for 14 days, followed by 7 days break in 21-day cycles throughout the study.

This multi-center trial will be conducted in the United States and Japan. The overall time to participate in this study is approximately 24 months. Participants will make multiple visits to the clinic. Participants in both Western cohort and disease specific cohorts will be followed for progression-free survival every 12 weeks after the last dose of the study drug until the occurrence of disease progression, loss to follow up, consent withdrawal, death, start of subsequent antineoplastic therapy, study termination, or until 6 months after discontinuation of the study treatment, whichever occurs first. Once disease progression is confirmed, participants in the disease-specific cohorts will be followed for overall survival every 12 weeks until death, loss to follow up, consent withdrawal, study termination, or transfer of a participant to a long term safety study, single participant investigational new drug application, or similar program after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female participants aged >=20 years (Japan) or >=18 years (United States).
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
3. Has pathologically confirmed metastatic pancreatic adenocarcinoma that has progressed after, at least, a first line of standard systemic chemotherapy for the metastatic disease, OR participants with pathologically confirmed metastatic adenocarcinoma of the colon or rectum who have progressed to at least 2 lines of standard systemic chemotherapy for the metastatic disease, OR participants with pathologically confirmed locally advanced or metastatic sqEC that has progressed after at least a first line of standard systemic therapy for metastatic disease. First-line participants can be enrolled if a platinum doublet is contraindicated or refused by the participants, OR pathologically confirmed locally advanced or metastatic sqNSCLC that has progressed after at least 2 lines of standard systemic therapy for metastatic disease.
4. For the Western safety cohort only: participants with locally advanced or metastatic solid tumor for whom no standard treatment with an established survival benefit is available or if the participant refuses other standard therapy.
5. For disease-specific cohort participants: measurable disease per RECIST v. 1.1
6. Left ventricular ejection fraction greater than (>) 50% as measured by ECHO or MUGA scan within 4 weeks before receiving the first dose of study drug.
7. Recovered to Grade 1 or baseline from all toxic effects of previous therapy (except alopecia or neuropathy).
8. Suitable venous access for the study-required blood sampling.
9. For the Western safety cohort only: willingness to undergo serial skin tissue biopsies.
10. For disease-specific cohort participants: Must have an archival (banked) tumor sample or agree to have a new (fresh) tumor biopsy during the screening period. If a new tumor sample is needed, the disease should be accessible for a nonsignificant risk biopsy procedure (those occurring outside the brain, lung/mediastinum, and pancreas, or obtained with endoscopic procedures not extending beyond the stomach or bowel). For participants in the Western safety cohort, this biopsy is optional.

Exclusion Criteria:

1. Participants who require continuous use of proton pump inhibitors (PPIs) or histamine-2 (H2) receptor antagonists and participants who are taking PPIs within 5 days before the first dose of study drug.
2. Treatment with clinically significant enzyme inducers, such as phenytoin, carbamazepine, phenobarbital, rifampin, rifabutin, rifapentine, or Saint John's wort within 14 days before the first dose of study drug.
3. Treatment with any systemic anticancer treatment (including investigational products) within 30 days or 5 half-lives, whichever is shorter, before the first dose of study drug.
4. History of any of the following within the last 3 months before administration of the first dose of study drug:

   * Ischemic myocardial event including angina requiring therapy and artery revascularization procedures, myocardial infarction, and unstable symptomatic ischemic heart disease.
   * Ischemic cerebrovascular event, including transient ischemic attack and artery, revascularization procedures.
   * Significant, uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation, or ventricular tachycardia).
   * New York Heart Association Class III to IV heart failure.
   * Any other cardiac condition that, in the opinion of the investigator, could pose an additional risk for participation in the study (example, pericardial effusion or restrictive cardiomyopathy).
   * Baseline prolongation of the QT interval corrected for heart rate (HR) using Fridericia's formula [QT interval corrected for heart rate using Fridericia's formula (QTcF); example, repeated demonstration of QTcF interval >480 millisecond (ms), history of congenital long QT syndrome, or torsades de pointes].
5. Hypertension that is unstable or not controlled by medication.
6. History of uncontrolled brain metastasis unless:

   * Previously treated with surgery, whole-brain radiation, or stereotactic radiosurgery, and
   * Stable disease (SD) for >=30 days, without steroid use (or stable steroid dose established for >=14 days before the first dose of TAK-931).
7. Known history of human immunodeficiency virus infection.
8. Known hepatitis B virus (HBV) surface antigen seropositive or detectable hepatitis C virus (HCV) infection viral load. Note: Participants who have positive HBV core antibody or HBV surface antigen antibody can be enrolled but must have an undetectable HBV viral load.
9. Prior treatment with radiation therapy involving >=25% of the hematopoietically active bone marrow within 3 months before the first dose of study drug.
10. Participants with known microsatellite instability-high (MSI-H) genotype or known wild type tumor protein 53 (TP53) per local testing.
11. Western Safety Cohort Only: Participants with Japanese heredity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (8):
  - Sarah Cannon Research Institute Oncology Research Consortium, Denver, Colorado
  - Sarah Cannon Research Institute, Sarasota, Florida
  - Allina Health Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - SCRI - Tennessee Oncology - Nashville - Southern Hills Clinic, Nashville, Tennessee
  - Virginia Mason Medical Center, Seattle, Washington
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in Japan and the United States from 25 October 2017 to 24 August 2020.
Pre-assignment Details: The study had two parts, Part 1 (Safety Cohort) enrolled western participants with locally advanced/metastatic solid tumors to receive TAK-931 and assessed safety, tolerability and pharmacokinetics. In Part 2, participants were enrolled into Tumor (Disease)-Specific Cohorts based on tumor criteria: pancreatic cancer, metastatic colorectal cancer (CRC), squamous esophageal cancer (sqEC), squamous non-small-cell lung cancer (sqNSCLC) to receive TAK-931 and were assessed for antitumor activity.
Period: Overall Study
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Started | 12 | 15 | 35 | 21 | 18
Completed | 0 | 2 | 5 | 0 | 1
Not Completed | 12 | 13 | 30 | 21 | 17
Not completed — Death | 10 | 13 | 17 | 12 | 8
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 1
Not completed — Site Terminated by Sponsor | 0 | 0 | 4 | 7 | 5
Not completed — Reason not Specified | 2 | 0 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort | Total
Number analyzed (Participants) | 12 | 15 | 35 | 21 | 18 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (7.16) | 63.1 (12.27) | 58.3 (11.93) | 64.2 (7.71) | 64.4 (7.74) | 61.5 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 19 | 4 | 7 | 40
  Male | 7 | 10 | 16 | 17 | 11 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 11 | 12 | 34 | 21 | 18 | 96
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 8 | 16 | 2 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 1 | 1 | 8
  White | 9 | 12 | 24 | 4 | 15 | 64
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 0 | 3 | 8 | 16 | 2 | 29
  United States | 12 | 12 | 27 | 5 | 16 | 72
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for height at the Baseline.
  cm
    number analyzed (Participants) | 12 | 15 | 34 | 20 | 18 | 99
    (all) | 172.47 (13.371) | 170.61 (11.596) | 168.64 (10.203) | 167.11 (7.975) | 172.26 (10.693) | 169.75 (10.513)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with data available for weight at the Baseline.
  kg
    number analyzed (Participants) | 12 | 15 | 35 | 20 | 18 | 100
    (all) | 79.33 (16.052) | 73.22 (22.763) | 79.90 (17.457) | 57.07 (10.358) | 77.70 (18.770) | 73.87 (19.076)
Substance Use [Count of Participants; unit: Participants] — Population: Data for substance use was collected only for sqEC and sqNSCLC cohorts. Number analyzed is the number of participants with data available for substance use at Baseline.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 20 | 18 | 38
    Tobacco | 0 | 0 | 0 | 12 | 3 | 15
    Cigarette | 0 | 0 | 0 | 6 | 15 | 21
    Cigar | 0 | 0 | 0 | 1 | 0 | 1
    Pipe | 0 | 0 | 0 | 1 | 0 | 1
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 12 | 15 | 35 | 2 | 1 | 65
  Current Smoker | 0 | 0 | 0 | 3 | 7 | 10
  Former Smoker | 0 | 0 | 0 | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLTs) in Western Safety Cohort
Description: DLT:Any following event related to TAK-931 assessed by Common Terminology Criteria for Adverse Events(CTCAE) version4.03;Non-febrile Grade 4 neutropenia; febrile neutropenia: Grade >=3 neutropenia; Grade4 thrombocytopenia; Grade >=3 thrombocytopenia of any duration accompanied by Grade 2 bleeding or requiring transfusion; delay in initiation of Cycle 2 by >14 days due to lack of adequate recovery of treatment-related hematological or nonhematologic toxicities; Grade 2 ejection fraction decreased by echocardiogram(ECHO) or multiple gated acquisition(MUGA) scan; Grade 4 laboratory abnormalities; other Grade 2 nonhematologic toxicities considered by investigator to be related to study drug and dose-limiting; Participants receiving <50% of doses (<7 doses) of planned TAK-931 dosing in Cycle 1 due to study drug-related adverse events(AEs); Grade >=3 nonhematologic toxicity with few exceptions: Grade 3 arthralgia/myalgia, fatigue, laboratory abnormalities, nausea and/or emesis or diarrhea.
Time Frame: Cycle 1 (each cycle = 21 days)
Population: DLT-evaluable Analysis Set included all participants in the Western Safety Cohort who received at least 1 of their planned TAK-931 doses during their first cycle of treatment (unless interrupted by related AEs) and who had sufficient follow-up data to allow the investigators and sponsor to determine whether a DLT occurred. As pre-specified in the protocol, DLTs were collected only from participants in the Western Safety Cohort who were evaluable in DLT-evaluable Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Western Safety Cohort
Number analyzed (Participants) | 2
percentage of participants | 50

2. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), TEAEs Leading to Dose Modifications and TEAEs Leading to Treatment Discontinuation in Western Safety Cohort
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an adverse event with an onset that occurred after receiving study drug. An SAE was any untoward medical occurrence or effect that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically important due to other reasons than the above mentioned criteria.
Time Frame: From first dose of the study drug up to 30 days after the last dose (Up to approximately 15 months)
Population: Safety Analysis Set included all participants who received any amount of study drug. As pre-specified in the protocol, this outcome measure reports data only in the participants with locally advanced or metastatic solid tumors in the Western Safety Cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Western Safety Cohort
Number analyzed (Participants) | 12
percentage of participants
  TEAEs | 100
  SAEs | 58.3
  TEAEs Leading to Dose Modifications | 33.3
  TEAEs Leading to Treatment Discontinuation | 8.3

3. Primary Outcome: Disease Control Rate (DCR) in Tumor-Specific Cohorts
Description: DCR was defined as percentage of participants documented to have unconfirmed CR, PR, or SD for at least 6 weeks from treatment initiation according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as the best response. CR was defined as disappearance of all lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of lesions, taking as reference the baseline sum LD. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started. PD was defined as at least a 20% increase in the sum of the LD of lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From first dose up to end of treatment (Up to approximately 14 months)
Population: Response-evaluable Analysis Set included all participants who received at least 1 dose of study drug, had measurable disease at Baseline, and had at least 1 post-baseline response assessment. As pre-specified in the protocol, this outcome measure evaluated and reported data for participants only in the Tumor-Specific Cohorts.
Measure: Number; unit: percentage of participants
Arm/Group | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 13 | 31 | 19 | 17
percentage of participants | 46.2 [26.4 to 66.9] | 51.6 [38.7 to 64.3] | 52.6 [35.8 to 69.0] | 58.8 [40.6 to 75.4]

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-931
Time Frame: Cycle 1 (each cycle = 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: Pharmacokinetic (PK) Analysis Set included all participants for whom there was sufficient dosing and TAK-931 concentration-time data to reliably estimate the PK parameters. As prespecified in the protocol, data for intensive PK sampling was collected only for participants in Western Safety Cohort, Pancreatic Cancer Cohort, and Metastatic CRC Cohort. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 12 | 15 | 34
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 12 | 12 | 13
  Cycle 1 Day 1 | 173.61 (59.677) | 204.69 (90.527) | 185.46 (61.158)
  Cycle 1 Day 8: number analyzed (Participants) | 12 | 10 | 11
  Cycle 1 Day 8 | 196.17 (73.702) | 180.55 (75.036) | 216.18 (121.488)

5. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-931
Time Frame: Cycle 1 (each cycle = 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: PK Analysis Set included all participants for whom there was sufficient dosing and TAK-931 concentration-time data to reliably estimate the PK parameters. As prespecified in the protocol, data for intensive PK sampling was collected only for participants in Western Safety Cohort, Pancreatic Cancer Cohort, and Metastatic CRC Cohort. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Median (Full Range); unit: hour
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 12 | 15 | 34
hour
  Cycle 1 Day 1: number analyzed (Participants) | 12 | 12 | 13
  Cycle 1 Day 1 | 1.57 [0.8 to 2.2] | 2.00 [0.5 to 6.3] | 1.85 [0.9 to 6.0]
  Cycle 1 Day 8: number analyzed (Participants) | 12 | 10 | 11
  Cycle 1 Day 8 | 1.59 [1.0 to 4.0] | 2.00 [1.0 to 4.3] | 1.97 [1.0 to 4.0]

6. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-931
Time Frame: Cycle 1 (each cycle = 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 12 | 15 | 34
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 12 | 12 | 13
  Cycle 1 Day 1 | 1190.22 (540.877) | 1166.40 (362.856) | 1302.40 (391.035)
  Cycle 1 Day 8: number analyzed (Participants) | 11 | 10 | 11
  Cycle 1 Day 8 | 1475.88 (749.707) | 1290.72 (615.542) | 1542.82 (507.733)

7. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-931
Time Frame: Cycle 1 (each cycle = 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 12 | 15 | 34
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 12 | 12 | 13
  Cycle 1 Day 1 | 1165.52 (552.287) | 1114.23 (388.844) | 1311.41 (388.557)
  Cycle 1 Day 8: number analyzed (Participants) | 12 | 10 | 11
  Cycle 1 Day 8 | 1426.70 (774.257) | 1289.33 (616.737) | 1551.57 (497.856)

8. Secondary Outcome: CLr: Renal Clearance of TAK-931
Description: CLr is a measure of apparent clearance of the drug from the plasma, renal clearance is a measure of drug excreted through kidneys/urine per unit time.
Time Frame: Cycle 1 (each cycle = 21 days) Day 1 pre-dose and at multiple timepoints (up to 8 hours urine sampling) post-dose
Population: PK Analysis Set included all participants for whom there was sufficient dosing and TAK-931 concentration-time data to reliably estimate the PK parameters. As prespecified in the protocol, data for urine PK sampling was collected only for participants in Western Safety Cohort. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Western Safety Cohort
Number analyzed (Participants) | 4
L/h | 2.16 (1.913)

9. Secondary Outcome: t1/2z: Terminal Disposition Phase Half-life for TAK-931
Time Frame: Cycle 1 (each cycle = 21 days) Day 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: PK Analysis Set included all participants for whom there was sufficient dosing and TAK-931 concentration-time data to reliably estimate the PK parameters. As prespecified in the protocol, data for intensive PK sampling was collected only for participants in Western Safety Cohort, Pancreatic Cancer Cohort, and Metastatic CRC Cohort. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Median (Full Range); unit: hour
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 11 | 10 | 11
hour | 5.95 [4.3 to 6.7] | 5.53 [3.7 to 8.0] | 6.18 [4.8 to 8.4]

10. Secondary Outcome: CLss/F: Steady-state Apparent Oral Clearance for TAK-931
Description: CL/F was defined as apparent clearance of the drug from the plasma, calculated as the drug dose divided by AUC.
Time Frame: Cycle 1 (each cycle = 21 days) Day 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 11 | 10 | 11
L/h | 39.71 (14.135) | 45.58 (18.877) | 35.57 (10.778)

11. Secondary Outcome: Rac(AUC): Accumulation Ratio Based on AUC Over the Dosing Interval (AUCτ) for TAK-931
Time Frame: Cycle 1 (each cycle = 21 days) Day 8 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort
Number analyzed (Participants) | 11 | 10 | 11
ratio | 1.27 (0.317) | 1.10 (0.299) | 1.12 (0.203)

12. Secondary Outcome: Overall Response Rate (CR and PR)
Description: Overall response rate was defined as percentage of participants documented to have unconfirmed CR or PR according to RECIST v1.1 as the best response. CR was defined as disappearance of all lesions, PR was defined as at least a 30% decrease in the sum of the LD of lesions, taking as reference the baseline sum LD.
Time Frame: From first dose up to end of treatment (Up to approximately 14 months)
Population: Response-evaluable Analysis Set included all participants who received at least 1 dose of study drug, had measurable disease at Baseline, and had at least 1 post-baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 12 | 13 | 31 | 19 | 17
percentage of participants | 8.3 [0.90 to 28.7] | 0 [0 to 16.2] | 0 [0 to 7.20] | 5.3 [0.60 to 19.0] | 0 [0 to 12.7]

13. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a CR or PR to the date of first documentation of tumor progression. Per RECIST V1.1, CR was defined as disappearance of all lesions, PR was defined as at least a 30% decrease in the sum of the LD of lesions, taking as reference the baseline sum LD. PD was defined as at least a 20% increase in the sum of the LD of lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From first documented response until disease progression or end of treatment, whichever occurs first (Up to 14 months)
Population: Response-evaluable Analysis Set included all participants who received at least 1 dose of study drug, had measurable disease at Baseline, and had at least 1 post-baseline response assessment. Only responders were to be analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 0
months | NA [NA to NA] — Data for median; upper and lower limits of confidence interval (CI) were not available as all responders were censored. |  |  | NA [NA to NA] — Data for median; upper and lower limits of CI were not available as all responders were censored. |

14. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose to the date of first documentation of PD (including clinical progression or clinical deterioration) or death due to any cause, whichever occurs first. Per RECIST V1.1, PD was defined as at least a 20% increase in the sum of the LD of lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From date of randomization until disease progression or death, whichever occurs first (Up to approximately 34 months)
Population: Safety Analysis Set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 12 | 15 | 35 | 21 | 18
months | 2.05 [1.31 to 5.09] | 1.31 [0.99 to 2.76] | 1.45 [1.35 to 2.56] | 3.02 [1.25 to 3.58] | 2.12 [1.28 to 3.25]

15. Secondary Outcome: Overall Survival (OS) in the Tumor-Specific Cohorts
Description: OS was defined as the time from the date of first dose of study drug to death due to any cause.
Time Frame: Up to approximately 43 months
Population: Safety Analysis Set included all participants who received any amount of study drug. Participants without documentation of death at the time of analysis were censored at the date last known to be alive. As pre-specified in the protocol, this outcome measure evaluated and reported data for participants only in the Tumor-Specific Cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 15 | 35 | 21 | 18
months | 4.67 [1.77 to 7.06] | 7.72 [5.68 to 11.96] | 8.61 [3.94 to 42.71] | NA [NA to NA] — The median, upper and lower limits of 95% confidence interval were not evaluable due to fewer number of participants with events.

16. Secondary Outcome: Percentage of Participants With Grade >=3 TEAEs, SAEs, TEAEs Leading to Dose Modifications, and TEAEs Leading to Treatment Discontinuation in Tumor-Specific Cohorts
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it did not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an adverse event with an onset that occurred after receiving study drug. TEAEs were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, where Grade 3: Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; Grade 4:Life-threatening consequences, urgent intervention indicated; Grade 5:Death related to AE. An SAE was any untoward medical occurrence or effect that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically important due to other reasons than the above mentioned criteria.
Time Frame: From first dose of the study drug up to 30 days after the last dose (Up to approximately 15 months)
Population: Safety Analysis Set included all participants who received any amount of study drug. As pre-specified in the protocol, this outcome measure evaluated and reported data for participants only in the Tumor-Specific Cohorts.
Measure: Number; unit: percentage of participants
Arm/Group | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 15 | 35 | 21 | 18
percentage of participants
  Grade >=3 TEAEs | 73.3 | 54.3 | 57.1 | 44.4
  SAEs | 40.0 | 22.9 | 23.8 | 16.7
  TEAEs Leading to Dose Modifications | 53.3 | 48.6 | 52.4 | 38.9
  TEAEs Leading to Treatment Discontinuation | 13.3 | 8.6 | 9.5 | 0

17. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Laboratory Values, Reported as Adverse Events in Tumor-Specific Cohorts
Description: Clinical laboratory tests included hematology, clinical chemistry and urinalysis. The investigator determined if the results were clinically significant. Only those categories were reported which are clinically significant at post Baseline.
Time Frame: From first dose of the study drug up to 30 days after the last dose (Up to approximately 15 months)
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 15 | 35 | 21 | 18
percentage of participants
  Neutrophil Count Decreased | 26.7 | 17.1 | 38.1 | 27.8
  White Blood Cell Count Decreased | 20.0 | 8.6 | 42.9 | 5.6
  Lymphocyte Count Decreased | 13.3 | 0 | 0 | 5.6
  Aspartate Aminotransferase Increased | 6.7 | 2.9 | 0 | 5.6
  Alanine Aminotransferase Increased | 6.7 | 0 | 0 | 5.6
  Blood Bilirubin Increased | 0 | 2.9 | 0 | 0
  Hepatic Enzyme Increased | 6.7 | 0 | 0 | 0
  Blood Creatinine Increased | 20.0 | 0 | 4.8 | 0
  Blood Creatinine Decreased | 6.7 | 0 | 0 | 0
  Blood Urea Increased | 6.7 | 0 | 0 | 0
  Blood Chloride Decreased | 6.7 | 0 | 0 | 0
  Blood Sodium Decreased | 0 | 2.9 | 0 | 0
  Platelet Count Decreased | 0 | 5.7 | 4.8 | 0
  Blood Alkaline Phosphatase Increased | 6.7 | 5.7 | 0 | 0
  Blood Uric Acid Increased | 6.7 | 0 | 0 | 0
  Blood Glucose Increased | 6.7 | 0 | 0 | 0
  Blood Albumin Decreased | 6.7 | 0 | 0 | 0
  Protein Total Decreased | 6.7 | 0 | 0 | 0
  Haematocrit Decreased | 6.7 | 0 | 0 | 0
  Red Blood Cell Count Decreased | 6.7 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Sign Measurements, Reported as Adverse Events in Tumor-Specific Cohorts
Description: Vital signs included assessments of systolic and diastolic blood pressure (BP), heart rate (HR), and body temperature. The investigator determined if the results were clinically significant. Only those categories were reported which are clinically significant at post Baseline.
Time Frame: From first dose of the study drug up to 30 days after the last dose (Up to approximately 15 months)
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
Number analyzed (Participants) | 15 | 35 | 21 | 18
percentage of participants
  Orthostatic Hypotension | 0 | 2.9 | 0 | 0
  Tachycardia | 0 | 5.7 | 0 | 0
  Bradycardia | 0 | 2.9 | 0 | 0
  Atrial Fibrillation | 0 | 2.9 | 0 | 0
  Increase in HR | 0 | 2.9 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to approximately 43 months; Serious and Other Adverse Events: From first dose of the study drug up to 30 days after the last dose (Up to approximately 15 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. A total of 67 deaths occurred in this study. Since all the information for death data could not be collected, not all deaths could be reported in all-cause mortality.
Arm/Group | Western Safety Cohort | Pancreatic Cancer Cohort | Metastatic CRC Cohort | sqEC Cohort | sqNSCLC Cohort
All-Cause Mortality (participants affected / at risk) | 10/12 | 13/15 | 17/35 | 12/21 | 8/18
Serious Adverse Events (participants affected / at risk) | 7/12 | 6/15 | 8/35 | 5/21 | 3/18
Other Adverse Events (participants affected / at risk) | 5/12 | 8/15 | 27/35 | 14/21 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Western Safety Cohort (N=12) | Pancreatic Cancer Cohort (N=15) | Metastatic CRC Cohort (N=35) | sqEC Cohort (N=21) | sqNSCLC Cohort (N=18)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Western Safety Cohort (N=12) | Pancreatic Cancer Cohort (N=15) | Metastatic CRC Cohort (N=35) | sqEC Cohort (N=21) | sqNSCLC Cohort (N=18)
Nausea (Gastrointestinal disorders) | 3 | 5 | 16 | 7 | 7
Vomiting (Gastrointestinal disorders) | 1 | 3 | 14 | 2 | 7
Constipation (Gastrointestinal disorders) | 2 | 2 | 6 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 6 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 2 | 4 | 6 | 5
White blood cell count decreased (Investigations) | 0 | 1 | 3 | 7 | 1
Ejection fraction decreased (Investigations) | 2 | 1 | 0 | 0 | 2
Weight decreased (Investigations) | 2 | 1 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 6 | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 5 | 3 | 2 | 2
Malaise (General disorders) | 1 | 0 | 3 | 2 | 0
Early satiety (General disorders) | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 3 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 3 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/5 | 1/5 | 0/19 | 0/4 | 0/4 — Number of participants at risk in each arm is based on the female population in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03261947/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT03261947/SAP_001.pdf